CLINICAL TRIAL: NCT07352176
Title: Study on the Effectiveness and Safety of Confocal Laser Endomicroscopy Combined With Ultrafine Cryoprobe for Biopsy Diagnosis of Pulmonary Lesions
Brief Title: Study on the Effectiveness and Safety of CLE Combined With Cryobiopsy for Diagnosis of Pulmonary Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CLE-Cryo
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Lesion; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diffuse- Conventional Group (Active Comparator): The Diffuse-Conventional Group used conventional cryobiopsy for lung lesions.
  Interventions: Other: Conventional cryobiopsy
- Diffuse- Combined Group (Experimental): The Diffuse-Combined Group used CLE combined with cryobiopsy for lung lesions
  Interventions: Other: Confocal laser endomicroscopy combined cryobiopsy
- Localized - Convention Group (Active Comparator): The Localized-Conventional Group used conventional cryobiopsy for lung lesions.
  Interventions: Other: Conventional cryobiopsy
- Localized - Combined Group (Experimental): The Localized-Combined Group used CLE combined with cryobiopsy for lung lesions
  Interventions: Other: Confocal laser endomicroscopy combined cryobiopsy

INTERVENTIONS:
Other: Confocal laser endomicroscopy combined cryobiopsy — Patients in the combined group will undergo CLT combined with cryobiopsy for lung lesions.
  Arms: Diffuse- Combined Group; Localized - Combined Group
Other: Conventional cryobiopsy — Patients in the conventional group will underg cryobiopsy for lung lesions.
  Arms: Diffuse- Conventional Group; Localized - Convention Group

SUMMARY:
Forty subjects meeting the inclusion and exclusion criteria were recruited at a single center and signed informed consent forms. Among them, 20 patients in the diffuse group and 20 patients in the localized group were randomly assigned to the conventional radial endobronchial ultrasound combined with cryobiopsy group (conventional group) and the confocal laser endomicroscopy combined with cryobiopsy group (combined group). During the operation, the operator manipulated the bronchoscope to reach the lesion. After confirming the arrival at the lesion using radial endobronchial ultrasound/confocal laser endomicroscopy, cryobiopsy was performed, and the size of the sample was recorded. CBCT scanning was conducted after cryobiopsy. If there was no hole-in-lesion image, cryobiopsy was performed again under CBCT guidance. CBCT scanning was performed after biopsy to determine whether there were any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old with lung lesions indicated by chest CT;
2. Preoperative CT indicates that the lung lesion to be biopsied has a bronchus leading to it;
3. Able to understand and voluntarily sign the written informed consent form. -

Exclusion Criteria:

1. Patients with contraindications to anesthesia or bronchoscopy;
2. Patients with uncorrectable coagulation disorders;
3. Patients who cannot discontinue therapeutic anticoagulants within an appropriate time interval before surgery;
4. Patients with severe liver or kidney dysfunction, mental illness, etc.;
5. Pregnant or lactating patients;
6. Patients without a clear histological or clinical diagnosis;
7. Subjects deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 7 days after procedure
  The Incidence of adverse events = (the number of adverse event / the number of procedures) * 100%

SECONDARY OUTCOMES:
Diagnostic yield | Immediately after the procedure
  The diagnostic yield = (the number of successful diagnoses / the number of completed biopsies) * 100%
Hole-in-lesion rate | During the procedure
  The rate of "hole-in-lesion" = (The number of cases with "hole-in-lesion" / The total number of cases that completed biopsy) * 100% The definition of "Hole-in-lesion": After cryobiopsy, a CBCT scan is performed, and the CBCT image shows the presence of a cavity within the lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong 510163, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kramer T, Wijmans L, de Bruin M, van Leeuwen T, Radonic T, Bonta P, Annema JT. Bronchoscopic needle-based confocal laser endomicroscopy (nCLE) as a real-time detection tool for peripheral lung cancer. Thorax. 2022 Apr;77(4):370-377. doi: 10.1136/thoraxjnl-2021-216885. Epub 2021 Jun 25. PMID 34172559
- [Background] Wellikoff AS, Holladay RC, Downie GH, Chaudoir CS, Brandi L, Turbat-Herrera EA. Comparison of in vivo probe-based confocal laser endomicroscopy with histopathology in lung cancer: A move toward optical biopsy. Respirology. 2015 Aug;20(6):967-74. doi: 10.1111/resp.12578. Epub 2015 Jun 19. PMID 26094505
- [Background] Sorokina A, Danilevskaya O, Averyanov A, Zabozlaev F, Sazonov D, Yarmus L, Lee HJ. Comparative study of ex vivo probe-based confocal laser endomicroscopy and light microscopy in lung cancer diagnostics. Respirology. 2014 Aug;19(6):907-13. doi: 10.1111/resp.12326. Epub 2014 Jun 9. PMID 24909555